CLINICAL TRIAL: NCT01040130
Title: Randomised, Double-blind, Placebo-controlled, 3-way Cross-over Study to Determine the Effect of Treatment of Orally Inhaled BI 1744 CL (5 µg [2 Actuations of 2.5 µg] and 10 µg [2 Actuations of 5 µg]) Delivered by the Respimat® Inhaler on Exercise Endurance Time During Constant Work Rate Cycle Ergometry in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Treatment BI 1744 CL (5 and 10 mcg) Versus Placebo on Exercise Endurance Time During Constant Work Rate Cycle Ergometry I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.37; 2009-014395-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol

ARMS (3):
- Olodaterol (BI 1744) Low (Experimental): Low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744); Drug: Olodaterol (BI 1744) Placebo
- Olodaterol (BI 1744) High (Experimental): High dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)
- Placebo (Placebo Comparator): Olodaterol (BI 1744) placebo inhaled once daily from the Respimat inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on exercise endurance time in COPD patients
  Arms: Olodaterol (BI 1744) High
Drug: Olodaterol (BI 1744) — Comparison of low and high doses on exercise endurance time in COPD patients
  Arms: Olodaterol (BI 1744) Low
Drug: Placebo — Comparison of low and high dose and placebo on exercise endurance time in COPD patients
  Arms: Placebo
Drug: Olodaterol (BI 1744) — Comparison of low and high dose
  Arms: Olodaterol (BI 1744) Low
Drug: Olodaterol (BI 1744) Placebo — Placebo that represents olodaterol
  Arms: Olodaterol (BI 1744) Low

SUMMARY:
To compare the effects of BI 1744 CL versus placebo on exercise tolerance after 6 weeks of treatment in patients with Chronic Obstructive Pulmonary Disease

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent prior to participation.
2. Diagnosis of chronic obstructive pulmonary disease and post-bronchodilator FEV1(Forced Expiratory Volume in 1 sec) <80% of predicted normal and post-bronchodilator FEV1(Forced Expiratory Volume in 1 sec)/FVC of < 70% at Visit 1.
3. Male or female between 40 and 75 years of age.
4. Current or ex-smokers with smoking history of more than 10-pack years.
5. Able to perform technically acceptable pulmonary function tests, multiple exercise tests and able to maintain records.
6. Able to inhale medication in a competent manner from a metered-dose inhaler and Respimat inhaler.

Exclusion criteria:

1. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an SGOT >x2 ULN, SGPT >x2 ULN, bilirubin >x2 ULN or creatinine >x2 ULN.
2. Patients with a history of asthma and/or total blood eosinophil count of 600 cells/mm3.
3. Patients with thyrotoxicosis, paroxysmal tachycardia (>100 beats per minute).
4. Patients with a history of myocardial infarction within 1 year of screening visit, unstable or life-threatening cardiac arrhythmia, hospitalization for heart failure within the past year, known active tuberculosis, a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years, life-threatening pulmonary obstruction, cystic fibrosis, clinically evident bronchiectasis, significant alcohol or drug abuse or contraindications to exercise.
5. Patients who have undergone thoracotomy with pulmonary resection.
6. Patients being treated with oral beta-adrenergics or oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
7. Patients who regularly use daytime oxygen for more than one hour per day.
8. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program.
9. Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea.
10. Pregnant or nursing women.
11. Women of childbearing potential not using two effective methods of birth control (one barrier and one non-barrier).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- Australia (4):
  - 1222.37.6171 Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - 1222.37.6174 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1222.37.6173 Boehringer Ingelheim Investigational Site, Heidelberg, Victoria
  - 1222.37.6172 Boehringer Ingelheim Investigational Site, Melbourne, Victoria
- Austria (2):
  - 1222.37.4371 Boehringer Ingelheim Investigational Site, Gänserndorf
  - 1222.37.4372 Boehringer Ingelheim Investigational Site, Neumarkt am Wallersee
- Canada (3):
  - 1222.37.1072 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1222.37.1074 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1222.37.1073 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
- France (6):
  - 1222.37.33005 Boehringer Ingelheim Investigational Site, Béthune
  - 1222.37.33002 Boehringer Ingelheim Investigational Site, Montpellier
  - 1222.37.33001 Boehringer Ingelheim Investigational Site, Nîmes
  - 1222.37.33006 Boehringer Ingelheim Investigational Site, Paris
  - 1222.37.33004 Boehringer Ingelheim Investigational Site, Perpignan
  - 1222.37.33003 Boehringer Ingelheim Investigational Site, Strasbourg
- Germany (4):
  - 1222.37.4970 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.37.4972 Boehringer Ingelheim Investigational Site, Halle
  - 1222.37.4973 Boehringer Ingelheim Investigational Site, Magdeburg
  - 1222.37.4971 Boehringer Ingelheim Investigational Site, Rüdersdorf

REFERENCES:
- [Derived] Maltais F, Kirsten AM, Hamilton A, De Sousa D, Voss F, Decramer M. Evaluation of the effects of olodaterol on exercise endurance in patients with chronic obstructive pulmonary disease: results from two 6-week crossover studies. Respir Res. 2016 Jul 6;17(1):77. doi: 10.1186/s12931-016-0389-5. PMID 27383762

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, double-blind, placebo-controlled, 3-way crossover trial. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Groups:
- Placebo / Olo 5mcg / Olo 10mcg: Patients were administered placebo in the first period, Olodaterol 5 mcg qd in the second period and Olodaterol 10 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Placebo / Olo 10mcg / Olo 5mcg: Patients were administered placebo in the first period, Olodaterol 10 mcg qd in the second period and Olodaterol 5 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg / Placebo / Olo 10mcg: Patients were administered Olodaterol 5 mcg qd in the first period, placebo in the second period and Olodaterol 10 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg / Olo 10mcg / Placebo: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 10 mcg qd in the second period and placebo in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg / Placebo / Olo 5mcg: Patients were administered Olodaterol 10 mcg qd in the first period, placebo in the second period and Olodaterol 5 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg / Olo 5mcg / Placebo: Patients were administered Olodaterol 10 mcg qd in the first period, Olodaterol 5 mcg qd in the second period and placebo in the third period. Olodaterol was administered via the Respimat inhaler.
Period: Overall Study
Arm/Group | Placebo / Olo 5mcg / Olo 10mcg | Placebo / Olo 10mcg / Olo 5mcg | Olo 5mcg / Placebo / Olo 10mcg | Olo 5mcg / Olo 10mcg / Placebo | Olo 10mcg / Placebo / Olo 5mcg | Olo 10mcg / Olo 5mcg / Placebo
Started | 25 (Number of patients entered and treated) | 25 | 25 | 25 | 25 | 26
Completed | 22 (Number of patients who did not discontinue from the trial.) | 22 | 23 | 20 | 25 | 22
Not Completed | 3 | 3 | 2 | 5 | 0 | 4
Not completed — Adverse Event | 1 | 1 | 0 | 5 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 1
Not completed — Other reasons not listed above | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Total: Total number of patients treated in the study. This was a randomised, double-blind, placebo-controlled, 3-way crossover trial. 151 patients were assigned randomly to one of 3 treatment sequences in which they received each of 3 treatments. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 116

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Endurance Time After 6 Weeks
Description: Primary endpoint was endurance time during constant work rate ergometry to symptom limitation at 75% of maximal work capacity after 6 weeks of treatment. Mixed effects model on log10 transformation data. Adjusted means are back transformed to report as geometric means. Standard errors (SEs) are calculated using the delta method.
Time Frame: 6 weeks
Population: Full analysis set (FAS). FAS is defined as all patients that were randomised, received treatment and had baseline data and any evaluable post-dose data for the primary endpoint.
Measure: Geometric Mean (Standard Error); unit: seconds
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 140 | 136
seconds | 369.81 (11.941) | 421.58 (13.459) | 420.72 (13.602)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline endurance time and period as fixed and patient as random effect. Means, CI back-transformed; Ratio to placebo = 1.140, 95% CI [1.065 to 1.221], Standard Error of Mean 0.040 — Olo 5 mcg divided by Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio to placebo = 1.138, 95% CI [1.062 to 1.219], Standard Error of Mean 0.040 — Olo 10 mcg divided by Placebo

2. Secondary Outcome: Adjusted Mean Inspiratory Capacity at Isotime After 6 Weeks
Description: Isotime is defined as the endurance time of the constant work rate exercise test of shortest duration from Baseline visit, and Week 6 of each of the three treatment periods.
Time Frame: 6 weeks
Population: Full analysis set (FAS). FAS is defined as all patients that were randomised, received treatment and had baseline data and any evaluable post-dose data for the primary endpoint. Only patients who have baseline and at least one post-baseline measurement available were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 140 | 135
liters | 1.917 (0.038) | 2.099 (0.038) | 2.091 (0.038)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.182, 95% CI [0.112 to 0.252], Standard Error of Mean 0.036 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.174, 95% CI [0.104 to 0.245], Standard Error of Mean 0.036 — Olo 10 mcg minus Placebo

3. Secondary Outcome: Adjusted Mean Borg Scale of Breathing Discomfort at Isotime After 6 Weeks
Description: Isotime is defined as the endurance time of the constant work rate exercise test of shortest duration from Baseline visit, and Week 6 of each of the three treatment periods.
  Borg scale rates discomfort with breathing at rest, during exercise and at end-exercise on a scale from 0=Nothing at all to 10=Maximal discomfort.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 140 | 136
Scores on a scale | 5.870 (0.185) | 5.104 (0.182) | 5.235 (0.185)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.766, 95% CI [-1.205 to -0.326], Standard Error of Mean 0.223 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.634, 95% CI [-1.077 to -0.192], Standard Error of Mean 0.225 — Olo 10 mcg minus Placebo

4. Secondary Outcome: Adjusted Mean Inspiratory Capacity at Pre-exercise After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 134 | 139 | 133
liters | 2.220 (0.032) | 2.478 (0.032) | 2.513 (0.032)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.258, 95% CI [0.191 to 0.325], Standard Error of Mean 0.034 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.294, 95% CI [0.226 to 0.362], Standard Error of Mean 0.035 — Olo 10 mcg minus Placebo

5. Secondary Outcome: Adjusted Mean Inspiratory Capacity at End of Exercise After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 140 | 135
liters | 1.887 (0.035) | 2.067 (0.035) | 2.024 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.180, 95% CI [0.107 to 0.252], Standard Error of Mean 0.037 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.137, 95% CI [0.064 to 0.210], Standard Error of Mean 0.037 — Olo 10 mcg minus Placebo

6. Secondary Outcome: Adjusted Mean Borg Scale of Breathing Discomfort at Pre-exercise After 6 Weeks
Description: Borg scale rates discomfort with breathing at rest, during exercise and at end-exercise on a scale from 0=Nothing at all to 10=Maximal discomfort.
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 140 | 135
Scores on a scale | 0.288 (0.041) | 0.185 (0.040) | 0.224 (0.041)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0447, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.103, 95% CI [-0.204 to -0.002], Standard Error of Mean 0.051 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.2132, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.064, 95% CI [-0.166 to 0.037], Standard Error of Mean 0.052 — Olo 10 mcg minus Placebo

7. Secondary Outcome: Adjusted Mean Borg Scale of Breathing Discomfort at End of Exercise After 6 Weeks
Description: as for outcome 6
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 140 | 136
Scores on a scale | 6.978 (0.143) | 6.890 (0.141) | 7.234 (0.143)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.5698, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.088, 95% CI [-0.391 to 0.216], Standard Error of Mean 0.154 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1003, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.256, 95% CI [-0.050 to 0.561], Standard Error of Mean 0.155 — Olo 10 mcg minus Placebo

8. Secondary Outcome: Adjusted Mean Functional Residual Capacity 30 Minutes Pre-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 134 | 139 | 134
liters | 4.977 (0.062) | 4.855 (0.061) | 4.862 (0.062)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0784, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.122, 95% CI [-0.258 to 0.014], Standard Error of Mean 0.069 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.1013, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.115, 95% CI [-0.252 to 0.023], Standard Error of Mean 0.070 — Olo 10 mcg minus Placebo

9. Secondary Outcome: Adjusted Mean Functional Residual Capacity 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 134 | 139 | 134
liters | 4.950 (0.064) | 4.740 (0.063) | 4.577 (0.064)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.210, 95% CI [-0.339 to -0.081], Standard Error of Mean 0.066 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.373, 95% CI [-0.503 to -0.243], Standard Error of Mean 0.066 — Olo 10 mcg minus Placebo

10. Secondary Outcome: Adjusted Mean Inspiratory Capacity 30 Minutes Pre-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 135 | 140 | 134
liters | 2.170 (0.040) | 2.289 (0.040) | 2.262 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.119, 95% CI [0.052 to 0.185], Standard Error of Mean 0.034 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0073, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.092, 95% CI [0.025 to 0.159], Standard Error of Mean 0.034 — Olo 10 mcg minus Placebo

11. Secondary Outcome: Adjusted Mean Inspiratory Capacity 1 Hour Post-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 135 | 140 | 134
liters | 2.221 (0.040) | 2.427 (0.040) | 2.437 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.206, 95% CI [0.136 to 0.275], Standard Error of Mean 0.035 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.216, 95% CI [0.146 to 0.285], Standard Error of Mean 0.036 — Olo 10 mcg minus Placebo

12. Secondary Outcome: Adjusted Mean Total Lung Capacity 30 Minutes Pre-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 135 | 140 | 134
liters | 7.142 (0.064) | 7.148 (0.063) | 7.121 (0.064)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.9239, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.006, 95% CI [-0.115 to 0.127], Standard Error of Mean 0.062 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.7368, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.021, 95% CI [-0.144 to 0.102], Standard Error of Mean 0.062 — Olo 10 mcg minus Placebo

13. Secondary Outcome: Adjusted Mean Total Lung Capacity 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 135 | 140 | 134
liters | 7.156 (0.066) | 7.142 (0.066) | 6.997 (0.067)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.8302, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.014, 95% CI [-0.146 to 0.118], Standard Error of Mean 0.067 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0202, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.159, 95% CI [-0.292 to -0.025], Standard Error of Mean 0.068 — Olo 10 mcg minus Placebo

14. Secondary Outcome: Adjusted Mean Forced Expiratory Volume in 1 Second, 30 Minutes Pre-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 137 | 137
liters | 1.475 (0.017) | 1.564 (0.017) | 1.576 (0.017)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.089, 95% CI [0.056 to 0.123], Standard Error of Mean 0.017 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.101, 95% CI [0.068 to 0.134], Standard Error of Mean 0.017 — Olo 10 mcg minus Placebo

15. Secondary Outcome: Adjusted Mean Forced Expiratory Volume in 1 Second, 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 137 | 137
liters | 1.473 (0.019) | 1.698 (0.019) | 1.699 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.224, 95% CI [0.191 to 0.258], Standard Error of Mean 0.017 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.226, 95% CI [0.193 to 0.259], Standard Error of Mean 0.017 — Olo 10 mcg minus Placebo

16. Secondary Outcome: Adjusted Mean Forced Vital Capacity, 30 Minutes Pre-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 135 | 136 | 136
liters | 3.212 (0.037) | 3.319 (0.037) | 3.310 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.107, 95% CI [0.046 to 0.167], Standard Error of Mean 0.031 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.098, 95% CI [0.037 to 0.158], Standard Error of Mean 0.031 — Olo 10 mcg minus Placebo

17. Secondary Outcome: Adjusted Mean Forced Vital Capacity, 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 135 | 136 | 136
liters | 3.187 (0.034) | 3.471 (0.034) | 3.477 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.285, 95% CI [0.227 to 0.342], Standard Error of Mean 0.029 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.290, 95% CI [0.233 to 0.348], Standard Error of Mean 0.029 — Olo 10 mcg minus Placebo

18. Secondary Outcome: Adjusted Mean Peak Expiratory Flow Rate, 30 Minutes Pre-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 137 | 137
liters/second | 4.374 (0.059) | 4.692 (0.059) | 4.677 (0.059)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.318, 95% CI [0.207 to 0.429], Standard Error of Mean 0.056 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.303, 95% CI [0.192 to 0.414], Standard Error of Mean 0.056 — Olo 10 mcg minus Placebo

19. Secondary Outcome: Adjusted Mean Peak Expiratory Flow Rate, 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 136 | 137 | 137
liters/second | 4.363 (0.063) | 4.949 (0.063) | 4.981 (0.063)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.585, 95% CI [0.470 to 0.701], Standard Error of Mean 0.063 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.618, 95% CI [0.502 to 0.734], Standard Error of Mean 0.059 — Olo 10 mcg minus Placebo

20. Secondary Outcome: Change From Baseline to Day 43 in Blood Pressure
Description: Change from Baseline to Day 43 in Blood Pressure with spirometry. Baseline is defined as mean of pre-treatment values at a given time point.
Time Frame: Baseline and Week 6
Population: Treated set. Statistics only include patients with both a baseline and a post dose value.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 131 | 133 | 136
mmHg
  Systolic blood pressure | -3.5 (15.64) | -2.7 (16.82) | -3.3 (16.47)
  Diastolic blood pressure | -1.7 (7.9) | -1.8 (8.36) | -1.1 (9.16)

21. Secondary Outcome: Change From Baseline to Day 43 in Pulse Rate
Description: Change from Baseline to Day 43 in Pulse rate with spirometry. Baseline is defined as mean of pre-treatment values at a given time point.
Time Frame: Baseline and Week 6
Population: Treated set. Statistics only include patients with both a baseline and a post dose value.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 138 | 142 | 141
beats/min | -5.1 (13.63) | -5.1 (13.88) | -3 (12.61)

22. Secondary Outcome: Number of Patients With Notable Changes in Heart Rate
Description: Number of Patients with notable changes in heart rate (HR). Notable HR increase defined as >=25% increase and on-treatment HR > 100 bpm; Notable HR decrease defined as >=25% decrease and on-treatment HR < 50 bpm.
Time Frame: Baseline and Week 6
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 138 | 141 | 140
percentage of participants
  30 min pre-dose: increase (N=138, 139, 140) | 0.7 | 0.7 | 0.7
  30 min pre-dose: decrease (N=138, 139, 140) | 1.4 | 2.9 | 2.1
  30 min pre-dose: no change (N=138, 139, 140) | 97.8 | 96.4 | 97.1
  40 min post-dose: increase (N=138, 141, 138) | 2.2 | 1.4 | 2.9
  40 min post-dose: decrease (N=138, 141, 138) | 4.3 | 5.0 | 6.5
  40 min post-dose: no change (N=138, 141, 138) | 93.5 | 93.6 | 90.6

23. Secondary Outcome: Number of Patients With Notable Increase in PR Intervals
Description: Number of Patients with notable increase in PR intervals. Notable PR interval increase defined as >=25% increase and on-treatment PR interval > 200 ms.
Time Frame: Baseline and Week 6
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 137 | 140 | 139
percentage of participants
  30 min pre-dose: increase (N=137, 137, 139) | 0.0 | 0.7 | 0.0
  30 min pre-dose: no increase (N=137, 137, 139) | 100.0 | 99.3 | 100.0
  40 min post-dose: increase (N=137, 140, 137) | 0.0 | 0.0 | 0.7
  40 min post-dose: no increase (N=137, 140, 137) | 100.0 | 100.0 | 99.3

24. Secondary Outcome: Number of Patients With Notable Increase in QRS Intervals
Description: Number of Patients with notable increase in QRS intervals. Notable QRS interval increase defined as >=10% increase and on-treatment QRS interval > 110 ms.
Time Frame: Baseline and Week 6
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 138 | 141 | 140
percentage of participants
  30 min pre-dose: increase (N=138, 139, 140) | 0.7 | 0.7 | 0.0
  30 min pre-dose: no increase (N=138, 139, 140) | 99.3 | 99.3 | 100.0
  40 min post-dose: increase (N=138, 141, 138) | 0.7 | 0.7 | 0.7
  40 min post-dose: no increase (N=138, 141, 138) | 99.3 | 99.3 | 99.3

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Serious Adverse Events (participants affected / at risk) | 3/143 | 3/147 | 3/143
Other Adverse Events (participants affected / at risk) | 8/143 | 10/147 | 5/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=143) | Olo 5 mcg (N=147) | Olo 10 mcg (N=143)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=143) | Olo 5 mcg (N=147) | Olo 10 mcg (N=143)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication